CLINICAL TRIAL: NCT05276700
Title: Alpha -1- Microglobulin (α1M) as an Early Biomarker in Renal Extrahepatic Manifestations of HCV-infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Safwat, principal investigator, Assiut University
Other Study IDs: α1M in HCV
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Renal Injury; HCV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case with hcv
- control without hcv

SUMMARY:
find the role of alpha one microglobulin (as an early renal tubular biomarker) to identify and evaluate the prevalence of early renal manifestations among patients with chronic HCV and compared these patients with HCV-negative healthy individuals

DETAILED DESCRIPTION:
Hepatitis C [HCV] infection is known to cause renal manifestations, which are discovered at a late stage when chronic kidney disease (CKD) has already occurred .

HCV is both a consequence and cause of renal impairment: first, dialysis patients have an increased risk of infection related to medical procedures and, second, HCV causes pathological changes to the kidneys .

HCV seems to influence both renal tubular and glomerular cells as described by different proteinuria profiles and hematuria findings. Tubular cell damage may be the earliest sign of renal dysfunction caused by HCV and could potentially be used to identify patients with risk for progression. Routine urine analysis could be used to identify high risk HCV patients for early treatment.

Identifying patients early is of paramount importance in order to offer a prompt intervention and to improve the prognosis in both settings, for this purposes, novel biomarkers could be used One promising biomarker is alpha-1-microglobulin (α1m), a low molecular weight glycosylated protein of molecular weight synthesized by hepatocytes, freely filtered across the glomerulus, and then reabsorbed by the proximal tubule . it can signal proximal tubule dysfunction: higher Uα1m concentrations indicate impaired tubular reabsorption . Small studies have previously shown that Uα1m concentrations increase in Acute kidney injury (AKI), reflect severity of AKI, and are associated with the need for dialysis after nonoliguric AKI . Elevated Uα1m correlates with interstitial fibrosis and tubular atrophy on kidney biopsy, representing chronic kidney damage . Furthermore, Uα1m appears to predict kidney function decline and CKD progression , Acute kidney injury risk and also associated with early tubulointerstitial renal diseases in HCV-glomerulopathy .

ELIGIBILITY:
Inclusion Criteria:

Hepatitis C virus (HCV )-positive patients: HCV Antibody and status confirmed by HCV-RNA positive who are either treatment naïve or previously treated.

3. HCV-negative control at outpatients.

Exclusion Criteria:

- 1. HIV-positive patients or Hepatitis B positive (HbsAg) patients or both. 2. Previous renal diseases. 3. Diabetes mellitus, Hypertension, Systemic Lupus erythematosus, Rheumatoid arthritis.

4. patients with Active malignancy. 5. Alcoholics.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 170 participants in 1:1 design (79 HCV positive patient were diagnosed as HCV positive by HCV+Abs and +ve real time PCR for HCV-RNA and 79 age and sex matched HCV negative as control, and fulfill the following inclusions criteria
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
to identify and evaluate the prevalence of early renal manifestations among patients with chronic HCV by using alpha one microglobulin (as an early renal tubular biomarker). | marsh 2022 - February 2024
  to identify and evaluate the prevalence of early renal manifestations among patients with chronic HCV by using alpha one microglobulin (as an early renal tubular biomarker).

CONTACTS AND LOCATIONS:
Overall Officials: Enas Alkareemy, Study Director — Assiut University

REFERENCES:
- [Background] Cacoub P, Comarmond C. Considering hepatitis C virus infection as a systemic disease. Semin Dial. 2019 Mar;32(2):99-107. doi: 10.1111/sdi.12758. Epub 2018 Dec 13. PMID 30549107
- [Background] Aguirre Valadez J, Garcia Juarez I, Rincon Pedrero R, Torre A. Management of chronic hepatitis C virus infection in patients with end-stage renal disease: a review. Ther Clin Risk Manag. 2015 Feb 27;11:329-38. doi: 10.2147/TCRM.S74282. eCollection 2015. PMID 25767389
- [Background] Kaartinen K, Vuoti S, Honkanen E, Loyttyniemi E, Singh R, Farkkila M. Tubular cell damage may be the earliest sign of renal extrahepatic manifestation caused by Hepatitis C. PLoS One. 2021 May 7;16(5):e0251392. doi: 10.1371/journal.pone.0251392. eCollection 2021. PMID 33961672
- [Background] Itoh Y, Kawai T. Human alpha 1-microglobulin: its measurement and clinical significance. J Clin Lab Anal. 1990;4(5):376-84. doi: 10.1002/jcla.1860040511. PMID 1700091
- [Background] Weber MH, Verwiebe R. Alpha 1-microglobulin (protein HC): features of a promising indicator of proximal tubular dysfunction. Eur J Clin Chem Clin Biochem. 1992 Oct;30(10):683-91. PMID 1283528
- [Background] Heise D, Rentsch K, Braeuer A, Friedrich M, Quintel M. Comparison of urinary neutrophil glucosaminidase-associated lipocalin, cystatin C, and alpha1-microglobulin for early detection of acute renal injury after cardiac surgery. Eur J Cardiothorac Surg. 2011 Jan;39(1):38-43. doi: 10.1016/j.ejcts.2010.05.044. Epub 2010 Jul 21. PMID 20650648
- [Background] Amer H, Lieske JC, Rule AD, Kremers WK, Larson TS, Franco Palacios CR, Stegall MD, Cosio FG. Urine high and low molecular weight proteins one-year post-kidney transplant: relationship to histology and graft survival. Am J Transplant. 2013 Mar;13(3):676-84. doi: 10.1111/ajt.12044. Epub 2013 Feb 15. PMID 23414180
- [Background] Bullen AL, Katz R, Lee AK, Anderson CAM, Cheung AK, Garimella PS, Jotwani V, Haley WE, Ishani A, Lash JP, Neyra JA, Punzi H, Rastogi A, Riessen E, Malhotra R, Parikh CR, Rocco MV, Wall BM, Bhatt UY, Shlipak MG, Ix JH, Estrella MM. The SPRINT trial suggests that markers of tubule cell function in the urine associate with risk of subsequent acute kidney injury while injury markers elevate after the injury. Kidney Int. 2019 Aug;96(2):470-479. doi: 10.1016/j.kint.2019.03.024. Epub 2019 May 7. PMID 31262489